CLINICAL TRIAL: NCT05872243
Title: A Prospective, Randomized, Double-blind, Controlled Trial of rTMS in the Treatment of Mild Alzheimer's Disease Guided by Personalized Brain Functional Sectors(pBFS)
Brief Title: pBFS Guided rTMS Treating Mild Alzheimer's Disease(AD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLXWAD2023
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Mild Alzheimer's Disease
Keywords: TMS, fMRI, AD, personalized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WMN group (Experimental): Active rTMS will be delivered to the tailored stimulation site within the working memory network.
  Interventions: Device: active rTMS
- DMN group (Experimental): Active rTMS will be delivered to the tailored stimulation site within the default mode network.
  Interventions: Device: active rTMS
- sham WMN group (Sham Comparator): Sham rTMS will be delivered to the tailored stimulation site within the working memory network.
  Interventions: Device: sham rTMS
- sham DMN group (Sham Comparator): Sham rTMS will be delivered to the tailored stimulation site within the default mode network.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active rTMS — Each participant will receive two 1800 pulse active rTMS in each session, with a 50-minute break in between. Participants will receive two separate sessions daily (a sum of 7200 pulses per day). The intervention will take place for 15 continuous days.
  Arms: DMN group; WMN group
Device: sham rTMS — Each participant will receive two 1800 pulse sham rTMS in each session, with a 50-minute break in between. Participants will receive two separate sessions daily (a sum of 7200 pulses per day). The intervention will take place for 15 continuous days.
  Arms: sham DMN group; sham WMN group

SUMMARY:
This study aims to investigate the effectiveness and safety of rTMS treatment under the guidance of personalized Brain Functional Sectors (pBFS) for the cognitive ability of patients with mild Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a neurodegenerative disorder characterized by memory impairment and cognitive decline. Personalized brain functional sectors (pBFS) using resting-state functional MRI scans have shown promise in precisely identifying individualized brain function networks. In this study, we aim to select tailored stimulation sites within the working memory network (WMN) or the default mode network (DMN) as intervention targets for mild AD patients using pBFS.

To evaluate the effectiveness and safety of this intervention, participants will be randomized into four groups: active repetitive transcranial magnetic stimulation (rTMS) to the WMN group, active rTMS to the DMN group, and sham rTMS to either the WMN or DMN group at a ratio of 2:2:1:1. Each participant will receive 3600 pulse active or sham rTMS in each session, consisting of two 1800 pulse treatments with a 50-minute break in between. Two separate treatment sessions will be administered daily, resulting in a sum of 7200 pulses per day. The intervention will be administered for 15 continuous days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (probable AD) based on the AD diagnostic criteria proposed by NIA-AA.
* Positive PET or positive cerebrospinal fluid test results for beta-amyloid (Aβ).
* Elementary school education or higher.
* MMSE scores between 20 and 26 (including 20 and 26), or 18 and 26 for those with elementary school education.
* Clinical Dementia Scale (CDR) score of 1, indicating mild dementia.
* Stable medication for Alzheimer's disease for at least 3 months prior to treatment.
* Availability of a reliable caregiver who can assist and accompany the patient throughout the study.
* Voluntary participation with signed informed consent by the patient or legal guardian.

Exclusion Criteria:

* Patients who have other causes of cognitive decline apart from AD, including but not limited to vascular dementia, Parkinson's disease dementia, dementia with Lewy bodies, frontotemporal dementia, and dementia due to endocrine system lesions or deficiencies of folic acid, vitamin B12 or other causes.
* Patients with significant focal lesions seen on MRI, including more than two infarct foci larger than 2 cm in diameter, infarct foci in key areas such as the thalamus, hippocampus, internal olfactory cortex, pars oligo-cortical, angular gyrus, cortical and other subcortical gray matter nuclei.
* Patients with moderate to severe cerebral white matter degeneration ( Fazekas score of 3-6).
* Patients unable to undergo TMS treatment or MRI scan due to metallic foreign bodies, implanted electronic devices, or claustrophobia.
* Patients with a history of seizures or epilepsy syndrome, or seizures within the past 12 months.
* Patients with acute cardiovascular and cerebrovascular events within the 3 months prior to screening.
* Patients with severe cardiac, pulmonary, hepatic, renal, and other systemic diseases that cannot be controlled with conventional medications.
* Patients with malignant tumors or a life expectancy of less than 1 year due to reasons other than AD.
* History of alcohol or drug abuse.
* Having received other TMS treatments within the past three months.
* Having participated, or is currently participating in other clinical trial programs within the past three months.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Post-treatment ADAS-Cog change | Pretreatment (baseline), Post-treatment (15 days)
  The Cognitive Subscale score change of the Alzheimer's Disease Assessment Scale, from baseline to post-treatment.

SECONDARY OUTCOMES:
Follow-up ADAS-Cog change | Pretreatment(baseline), follow-up (90 days)
  The Cognitive Subscale score change of the Alzheimer's Disease Assessment Scale, from baseline to follow-up
MMSE change | Pretreatment(baseline), post-treatment(15 days), follow-up (90 days)
  Change in Mini-Mental State Examination (MMSE) scores at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).

OTHER OUTCOMES:
MoCA change | Pretreatment(baseline), post-treatment (15 days), follow-up (90 days)
  Change in Montreal Cognitive Assessment (MoCA) scores at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).
NPI change | Pretreatment(baseline), post-treatment (15 days), follow-up (90 days)
  Change in Neuropsychiatric Inventory scores at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).
AVLT change | Pretreatment(baseline), post-treatment (15 days), follow-up (90 days)
  Change in Auditory Verbal Learning Test (AVLT) at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).
TMT change | Pretreatment(baseline), post-treatment (15 days), follow-up (90 days)
  Change in Trail Making Test (TMT)at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).
Digit span change | Pretreatment(baseline), post-treatment (15 days), follow-up (90 days)
  Change in Digit span at post-treatment (15 days) and follow-up (90 days) compared to baseline assessment (0 days).

CONTACTS AND LOCATIONS:
Overall Officials: HeSheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China